CLINICAL TRIAL: NCT06924281
Title: Team Science to Identify & Intervene on Metabolism- & Alcohol-Associated Liver Disease
Brief Title: Team Science (The Liver Health Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00000611; P20GM130414-06S1 (NIH)
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-09

CONDITIONS: Steatotic Liver Disease of Mixed Origin (MetALD)
Keywords: Metabolism and alcohol-associated liver disease; Motivational interviewing; Personalized feedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Intervention (Active Comparator): Participants randomly assigned to this arm will receive psychotherapy utilizing manualized principles of motivational interviewing with standard health information.
  Interventions: Behavioral: Brief motivational interviewing with standard health information
- Enhanced Intervention (Experimental): Participants randomly assigned to this arm will receive psychotherapy utilizing manualized principles of motivational interviewing that incorporates personalized feedback on self-reported alcohol intake and two scores from Fibroscan® liver imaging that indicate steatosis (liver fat) and fibrosis (liver scaring).
  Interventions: Behavioral: Brief motivational interviewing with personalized feedback

INTERVENTIONS:
Behavioral: Brief motivational interviewing with personalized feedback — The manualized intervention is delivered individually in two phases by an interventionist trained in motivational interviewing. The intervention includes liver health information and explains connections with weight-related behaviors. The enhanced (experimental) group receives personalized feedback, i.e., a summary of self-reported drinking patterns and results of liver imaging with Fibroscan®, i.e., steatosis (liver fat) and fibrosis (liver scaring) scores. The feedback is used to develop discrepancies between a goal of halting or reversing health risks associated with consuming alcohol versus continuing to drink. The sessions are matched in duration and interventionist skill level with the standard (control) group.
  Arms: Enhanced Intervention
Behavioral: Brief motivational interviewing with standard health information — The manualized intervention is delivered individually in two phases by an interventionist trained in motivational interviewing. The intervention includes liver health information and explains connections with weight-related behaviors. The standard (control) group does not receive personalized feedback. The sessions are matched in duration and interventionist skill level with the enhanced (experimental) group.
  Arms: Standard Intervention

SUMMARY:
Liver damage from alcohol intake and weight-related behaviors is preventable and treatable only through lifestyle changes. This mixed-methods randomized controlled trial compares standard and enhanced approaches to screening, brief intervention, and referral to treatment/prevention (SBIRT/P) to identify and intervene for metabolism- and alcohol-associated liver disease (MetALD). Our multidisciplinary team aims to show that integrating results of noninvasive liver screening with Fibroscan®, a painless ultrasound that measures stiffness and fat in the liver, can optimize our brief intervention. The study population is adults age 21+ who speak Spanish or English from underresourced communities with alcohol- and weight-related risks for MetALD.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age.
* Exceed alcohol intake screening guidelines for MetALD.
* Have a Body Mass Index (BMI) >=25 kg/m2.
* Be able to speak and read English or Spanish to provide written informed consent and understand written and oral instructions in English or Spanish.

Exclusion Criteria:

* Pre-existing liver disease or hepatocellular carcinoma or prior liver transplant.
* Pre-existing medical conditions that, in the opinion of the investigative team, would interfere with research participation (e.g., loss of kidney function, uncontrolled infections, multiorgan failure, uncontrolled upper gastrointestinal bleeding, other active malignancies except skin cancer).
* Pre-existing mental health conditions that, in the opinion of the investigative team, would interfere with the ability to provide informed consent and understand written and oral instructions (e.g., hepatic encephalopathy, psychotic disorder diagnosis or symptoms).
* Current pregnancy.
* Be anyone who, based on self-reported withdrawal symptoms and the opinion of the investigative team, could not currently safely be withdrawn from alcohol without medical detoxification.
* Currently receiving formalized psychosocial treatment for an alcohol use or drug problem and/or newly taking medications for an alcohol use or drug problem.
* Currently receiving formalized behavioral weight management treatment and/or newly taking weight loss medications.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Esperanza Hope Clinic, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Intervention | Enhanced Intervention
Started | 6 | 8
Completed | 5 | 7
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Intervention | Enhanced Intervention | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13) | 44 (17) | 43 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
High Body Mass Index Stratification Group [Count of Participants; unit: Participants] | 3 | 2 | 5
High Alcohol Consumption Level Stratification Group [Count of Participants; unit: Participants] | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion Screened With Alcohol Intake and Weight-related Risks for Metabolism and Alcohol-associated Liver Disease
Description: The primary feasibility outcome is the proportion screened who have alcohol intake and weight-related risks for metabolism and alcohol-associated liver disease. Alcohol intake risk is identified by the 3-item Alcohol Use Disorder Identification Test-Consumption subscale (AUDIT-C). Weight-related risk is identified by body mass index, calculated from weight and height.
Time Frame: Screening
Population: This is the number of participants who were identified by electronic health record reviews who responded to pre-screening questions.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-randomization Screening Phase: Arm/group is not applicable for this primary outcome measure, as screening occurred prior to randomization to standard/enhanced intervention groups.
Arm/Group | Pre-randomization Screening Phase
Number analyzed (Participants) | 58
Participants | 26

2. Primary Outcome: Proportion Eligible and Invited to Participate Who Agree to Noninvasive Liver Imaging With Fibroscan® and Arrive for Scheduled Baseline Appointment
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-randomization Screening Phase
Number analyzed (Participants) | 17
Participants | 14

3. Primary Outcome: Satisfaction With Fibroscan® Liver Imaging
Description: Satisfaction with liver screening is assessed with a single-item visual analog scale with 0 indicating low satisfaction and 100 indicating high satisfaction.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Intervention | Enhanced Intervention
Number analyzed (Participants) | 6 | 8
units on a scale | 88.5 (11.2) | 93.9 (7.1)

4. Secondary Outcome: Alcohol Intake Assessed by Timeline Followback Interview Before and After Intervention
Description: Timeline followback interviews will be individually administered in a semi-structured format by outcomes assessors who are masked to intervention condition. Interviews follow standardized procedures using a 30-day calendar to identify anchoring events, abstinent days, and types of alcohol consumed including ounces and alcohol by volume.
Time Frame: 30 days prior to intervention and 30 days after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Standard Intervention | Enhanced Intervention
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT06924281/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT06924281/SAP_001.pdf
  • Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT06924281/ICF_002.pdf